CLINICAL TRIAL: NCT06515340
Title: Effect of Allulose on Diet-induced Thermogenesis, Substrate Oxidation, Glycemic Response, and Satiety in Normal Weight Adults
Brief Title: Effect of Allulose on Diet-induced Thermogenesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Anderson Advanced Ingredients (Industry)
Responsible Party: Principal Investigator, Nick Bellissimo, PhD, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REB 2023-206 (A)
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Diet Induced Thermogenesis
Keywords: Adults; Allulose; Energy expenditure; Blood glucose; Appetite

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Allulose Dose 1 (Experimental): Treatment
  Interventions: Other: Allulose Dose 1
- Allulose Dose 2 (Experimental): Treatment
  Interventions: Other: Allulose Dose 2
- Allulose Dose 3 (Experimental): Treatment
  Interventions: Other: Allulose Dose 3

INTERVENTIONS:
Other: Allulose Dose 1 — 5 gram consumed orally
  Arms: Allulose Dose 1
Other: Allulose Dose 2 — 10 gram consumed orally
  Arms: Allulose Dose 2
Other: Allulose Dose 3 — 20 gram consumed orally
  Arms: Allulose Dose 3

SUMMARY:
The objective of this study is to investigate the dose-response effect of allulose on diet-induced thermogenesis, substrate oxidation, glycemic response, and subjective appetite in healthy normal weight adults.

DETAILED DESCRIPTION:
A within-subject, repeated measures, randomized, repeated measures design will be used. Participants (n= 10, 5 males, 5 females) will consume, in a random order, one of three varying doses of test treatments (allulose (5g), allulose (10g) or allulose (20g)) on 3 separate days. After treatment consumption, energy expenditure measurements via indirect calorimetry will be collected in 30-min interval (30-min measurement, 30-min rest) for 3 hours. Blood glucose will be measured at baseline and continuously for 3 hours via the Dexcom G6 continuous glucose monitoring system. Subjective appetite (hunger, fullness, desire to eat, prospective food consumption) will be measured via visual analogue scales at baseline and at the end of each energy expenditure measurement interval over 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Participants (18 - 45 years) who are considered healthy, are non-smokers, and have a body mass index (BMI) between 20 and 24.9 kg/m2 [World Health Organization classification of normal weight BMI].

Exclusion Criteria:

* Participants who have a fasting plasma glucose > 5.5 mmol/L indicative of impaired fasting glucose, previously diagnosed diabetes, known or uncertain pregnancy status at the screening visit, gastrointestinal disease, liver or kidney disease, have undergone a major medical or surgical event within the past 6 months, were or are on a diet, skip breakfast, smoke or have taken medication which would be a potential confounder with effects on metabolic and intake regulation.
* Those unable to complete the testing protocols or are intolerant or allergic to test-day ingredients.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Diet-induced thermogenesis | Collected at baseline (before treatment consumption) and 30-min intervals for 3 hours post-treatment consumption.
  Before treatment consumption, participants will be rested in a supine position for 30 min to reach a steady resting state in an isolated, dimly lit room under controlled temperature and humidity conditions. Resting energy expenditure (REE) will be determined by indirect calorimetry (ParvoMedics TrueOne2400 automated metabolic gas analysis system, ParvoMedics, Sandy, UT, USA) under a ventilated hood for 30 min. Post-treatment consumption, respiratory gases will be measured in 30 min intervals for 3 hours under the ventilated hood using the indirect calorimeter, with a 30 min rest break between measurements. Diet-induced thermogenesis (kcal/h) will be calculated as the increase in energy expenditure above baseline REE over the duration of the measurements.

SECONDARY OUTCOMES:
Substrate oxidation | Collected at baseline (before treatment consumption) and 30-min intervals for 3 hours post-treatment consumption.
  During the assessment of diet-induced thermogenesis via indirect calorimetry, respiratory exchange ratio will be monitored to assess the effects on substrate utilization. Energy expenditure and substrate oxidation rates for each hourly interval will be calculated using average VO2 and VCO2 measurements.
Glycemic response | Collected at baseline (before treatment consumption) and 5-min intervals for 3 hours post-treatment consumption.
  Blood glucose concentrations will be collected using the Dexcom Continuous Glucose Monitoring system, which collects glucose measurements from the interstitial fluid. The sensor will provide blood glucose data every five minutes which will be used to evaluate glycemic response over the duration of each session. Continuous glucose monitors will be inserted by the participants on their abdomen following the manufacturer instructions and with the assistance of a trained research assistant.
Subjective appetite | Collected at baseline (before treatment consumption) and 30 min intervals for 3 hours post-treatment consumption.
  Measured using visual analogue scales (VAS). Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings. Questions will include desire to eat, fullness, hunger, and prospective food consumption. Individual questions will be used to form a composite score.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Centre for Urban Innovation (CUI-109), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No